CLINICAL TRIAL: NCT01112189
Title: Postoperative Lymphedema Treatment in Upper Extremities Following Axillary Lymphadenectomy by Transplanting Autologous Endothelial Progenitor Cells (EPC)
Brief Title: Use of Stem Cells in Lymphedema Post Mastectomy
Acronym: SCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Dr. med Gerardo Enrique Muñoz Maldonado, Hospital Universitario "Dr. José Eleuterio González"
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CG08-005
Record Dates: First submitted 2010-04-20; First posted 2010-04-28 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2010-02

CONDITIONS: Lymphedema; Breast Cancer
Keywords: Lymphedema; Stem cells; Mastectomy; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with stem cells (Experimental): Patients that receive the stem cells treatment
  Interventions: Procedure: Autologous transplant
- Compressed sleeve treatment (Active Comparator): Patients that will receive the compressed sleeve treatment
  Interventions: Other: Compressed sleeve treatment

INTERVENTIONS:
Procedure: Autologous transplant — Patients will be stimulated 3 days with Filgrastrim 300 micrograms per day. On the 4th day the autologous transplant of stem cells will be performed.
  Other Names: Stem Cells transplant
  Arms: Patients with stem cells
Other: Compressed sleeve treatment — Week 1-2: With compressed sleeve treatment.
  Week 3 -4: Without treatment.
  Week 5 - 6: With compressed sleeve treatment
  Other Names: Compressive sleeve treatment
  Arms: Compressed sleeve treatment

SUMMARY:
The post-mastectomy lymphedema is a complication of removal of the breast and nodal plexus that causes accumulation of lymph and subsequent enlargement of the upper limb. It is the most common complication of all attributable to mastectomy with axillary dissection and which occurs in one third of patients who undergo radical mastectomy and radiotherapy post-operation. Currently the treatment of lymphedema of the upper limb is mainly the use of compression stockings, the use of pneumatic compression pumps and physiotherapy.

Multiple reports indicate that endothelial progenitor cells (EPC) can differentiate into various cell lines, reproduced and participate in neoangiogenesis. This study was conducted in the General Surgery Service, of the Hospital Universitario "Dr. José Eleuterio González "and proposes the EPC obtained autologous transplantation of bone marrow for the treatment of postoperative lymphedema in upper limb following axillary lymphadenectomy through the stimulation of lymphatic neoangiogenesis. The investigators studied 20 female patients over 18 years after axillary lymphadenectomy. The objective is to develop an innovative and definitive treatment for these patients and to analyze the costs and complications that this treatment may have.

DETAILED DESCRIPTION:
Phase 1:

The procedure will be as follows:

10 patients were recruited in the General Surgery or Oncology meeting the inclusion criteria. During the study, patients can´t use any other kind of treatment for the lymphedema.

Visit 1: We explain the procedure by inviting patients to participate after signing informed consent. There will be a complete medical history, review of inclusion and exclusion criteria, signing a letter of informed consent, be requested general laboratory tests (blood count, biochemical profile), tele-ray.

Visit 2: Initiation colony stimulating factor (Filgrastim SC) to 300 micrograms per day for 3 consecutive days.

Visit 3: Conduct a puncture and bone marrow harvesting under local anesthesia of the posterior iliac crest with Jamshidi needle to aspirate (approximately 50 - 100ml). The product obtained will be centrifuged in a refrigerated centrifuge at 3500 Sigma EK15 ® rpm/15 minutes to 8 ° C with HES 6% (pentastarch 6g/100ml) to obtain the mononuclear cell layer. Once the cells were obtained will be transported to the operating room to manage the patient by intramuscular injection of 0.5 to 1 ml in 30 to 50 sites of the affected limb with a depth of about one centimeter, using a needle number 25. The administration will take place in the operating room under local anesthesia or sedation if necessary.

Visit 4 and subsequent: clinical evaluation will be conducted each week, especially data monitoring of infection in the puncture sites. At week 12 post-cell infusion, the latest revision will be made and carried out measurements in both arms to conclude and determine the outcome of treatment.

Phase 2 (Control group):

Another 10 patients with lymphedema will be included in a 6 week study to compare the most common treatment of the lymphedema, the compressed sleeves.

Visit 1: A complete medical history will be performed. A compression sleeve will be given to the patients for their use during the next 2 weeks.

Visit 2 and 3: On week 2 and 3 of the compression sleeve treatment, the patients will be measured in both upper extremities as well as assess the symptoms or not that patients present.

Visit 4 and 5: Patients will stop using the compression sleeve treatment for the next 2 weeks measured both upper extremities and interrogate patients about symptoms during this period.

Visit 6 and 7: The last 2 weeks of the study patients will be asked to restart the compressed sleeves treatment and measured both upper extremities and interrogate patients about symptoms presented during this stage of the study.

ELIGIBILITY:
Inclusion criteria:

* Patients with postsurgical lymphedema in upper extremities following axillary lymphadenectomy.
* Female gender.
* Age over 18 years.
* Patients who wish to participate in the study.
* Informed consent signed.

Exclusion criteria:

* Patients with hypercoagulable states.
* Patients with a history of obstructive vascular disease in the brain, kidneys or heart.
* Patients with congestive heart failure (ejection fraction less than 30%)
* Active infectious process, serious, anywhere in the body.
* Patients over 75 years of age.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determine if the stem cells are effective in patients with lymphedema with the decreased of the volume of the affected limb and improvement of the symptomatology. | 3 months
  Patients will be measured in 4 different areas of both arms with a tape measure, before the transplant and weekly after the transplant for 3 months.
  Measure 1: 10 cm over the epicondyle. Measure 2: 5 cm over the the epicondyle. Measure 3: 5 cm under the the epicondyle. Measure 4: 15 cm under the the epicondyle Also a questionnaire of the most common symptoms will be given to the patients to mark their own symptoms before the transplant and 3 months after the transplant.

SECONDARY OUTCOMES:
Participants with Adverse Events as a Measure of Safety and Tolerability. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo E. Muñoz Maldonado, MD, Principal Investigator — Hospital Universitario Dr Jose Eleuterio Gonzalez
Locations (1):
- Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Thomas-MacLean R, Miedema B, Tatemichi SR. Breast cancer-related lymphedema: women's experiences with an underestimated condition. Can Fam Physician. 2005 Feb;51(2):246-7. PMID 16926934
- [Background] Levine M; Steering Committee on Clinical Practice Guidelines for the Care and Treatment of Breast Cancer. Clinical practice guidelines for the care and treatment of breast cancer: adjuvant systemic therapy for node-positive breast cancer (summary of the 2001 update). The Steering Committee on Clinical Practice Guidelines for the Care and Treatment of Breast Cancer. CMAJ. 2001 Mar 6;164(5):644-6. No abstract available. PMID 11258212
- [Background] Bumpers HL, Best IM, Norman D, Weaver WL. Debilitating lymphedema of the upper extremity after treatment of breast cancer. Am J Clin Oncol. 2002 Aug;25(4):365-7. doi: 10.1097/00000421-200208000-00009. PMID 12151966
- [Background] Kim H, Dumont DJ. Molecular mechanisms in lymphangiogenesis: model systems and implications in human disease. Clin Genet. 2003 Oct;64(4):282-92. doi: 10.1034/j.1399-0004.2003.00152.x. PMID 12974730
- [Derived] Maldonado GE, Perez CA, Covarrubias EE, Cabriales SA, Leyva LA, Perez JC, Almaguer DG. Autologous stem cells for the treatment of post-mastectomy lymphedema: a pilot study. Cytotherapy. 2011 Nov;13(10):1249-55. doi: 10.3109/14653249.2011.594791. PMID 21999374